CLINICAL TRIAL: NCT05426018
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Trial Evaluate the Efficacy and Safety of Oral Administration of Different Doses of SY-009 Capsule in Patients With T2DM for 12 Weeks
Brief Title: The Efficacy and Safety of Different Doses of SY-009 in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY009003
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
Keywords: Sodium glucose cotransporter-1 (SGLT-1) inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SY-009 -1 (Experimental): 0.5mg tid
  Interventions: Drug: SY-009 capsules
- SY-009-2 (Experimental): 1.0mg tid
  Interventions: Drug: SY-009 capsules
- SY-009-3 (Experimental): 1.5mg tid
  Interventions: Drug: SY-009 capsules
- Placebo (Placebo Comparator): tid
  Interventions: Drug: SY-009 capsules

INTERVENTIONS:
Drug: SY-009 capsules — 3 capsules each time (3 test drugs), 3 times a day (oral administration before breakfast, lunch, dinner or with meals)

SUMMARY:
SY-009 is a novel compound that inhibits sodium glucose cotransporter-1 (SGLT-1). The preclinical and phase 1 clinical trial data support to carry out phase II clinical trial in diabetes subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects were ≥ 18 years old and ≤ 75 years old at the first screening (visit 1);
2. At the first screening (visit 1) and the baseline period (visit 3), male weight ≥ 50kg, female weight ≥ 45kg, and body mass index (BMI) between 18.0 and 35.0 kg/m2 (including the critical value);
3. At the first screening (visit 1), the subjects had been diagnosed with type 2 diabetes for at least 3 months according to the WHO diagnostic criteria and classification in 1999;
4. The subjects had been receiving diet control and exercise therapy for 3 months before the first screening (visit 1), and had not received systematic treatment for diabetes during this period (the cumulative use of hypoglycemic drugs in recent 3 months was not more than 2 weeks, and no hypoglycemic drugs were used in recent 1 month);
5. The subjects' HbA1c at the first screening (visit 1) was between 7.5% and 10.5% (including the critical value); During the baseline period (visit 3), HbA1c was between 7.0% and 10.5% (including the critical value);
6. Subjects' fasting blood glucose ≤ 13.3mmol/l in the baseline period (visit 3);
7. Before the trial, the nature, significance, possible benefits, possible inconvenience, potential risks and discomfort of the trial have been understood in detail, and they have volunteered to participate in the clinical trial. They can communicate well with researchers, comply with the requirements of the whole trial, and have signed a written informed consent.

Exclusion Criteria:

1. Known allergic to the test drug (including the excipients of the test drug) or its analogues, or allergic constitution (such as allergic to two or more drugs, food and pollen), or having taken SGLT-1 or sglt-2 inhibitors in the past 1 year;
2. Received long-term (>2 weeks) systemic glucocorticoid therapy (excluding topical, ophthalmic or inhaled preparations) within 3 months before screening;
3. Diagnosed as type 1 diabetes, or gestational diabetes, or other special types of diabetes;
4. There is sufficient evidence of active diabetes proliferative retinopathy;
5. History of severe hypoglycemia (such as consciousness disorder and coma caused by hypoglycemia), or history of serious unconscious hypoglycemia;
6. History of acute metabolic complications of diabetes within 6 months before screening (diabetes ketoacidosis, hypertonic non ketoacidosis coma, diabetes lactic acidosis);
7. Serious trauma, serious infection or operation that may affect blood glucose control occurred within 1 month before screening;
8. There are obvious blood system diseases (such as aplastic anemia, myelodysplastic syndrome), or any disease that causes hemolysis or red blood cell instability (such as malaria), or hemoglobinopathy that may affect the determination of HbA1c level (such as sickle cell disease);
9. Have obvious autonomic neuropathy, such as urinary retention, postural hypotension, diabetes diarrhea or gastroparesis；
10. Habitual diarrhea, irritable bowel syndrome, clinically significant abnormal gastric emptying (such as gastric outlet obstruction), severe chronic gastrointestinal diseases (such as active ulcer within 6 months) or gastrointestinal surgery within 3 months before screening;
11. History of organ transplantation (excluding corneal transplantation), or other acquired or congenital immune system diseases, or clinically significant peripheral vascular diseases;
12. History of heart failure (NYHA grade III and IV), or history of acute myocardial infarction or unstable angina pectoris within 6 months before screening; Or have a history of coronary angioplasty, coronary stent implantation or coronary artery bypass surgery within 6 months before screening or have a recent cardiac surgery plan;
13. In the screening period, when no pacemaker was installed, grade II or III atrioventricular block or qtcb interval was prolonged >500 MS in 12 lead ECG;
14. Patients with abnormal thyroid function (such as thiourea and thyroid hormone drugs) whose treatment dose was not stable within the first 6 months were screened; Hypothyroidism with poor control or history of hypothyroidism;
15. Unstable weight (weight change more than 5kg) within 2 months before screening, or used drugs with weight control effect or performed surgery that can lead to unstable weight, or is currently in the weight loss plan and is not in the maintenance stage;
16. Poor blood pressure control (systolic blood pressure (SBP) ≥ 160mmhg and / or diastolic blood pressure (DBP) ≥ 100 mmHg);
17. At the first screening (visit 1), the subjects were positive for HBsAg, HCV antibody, Treponema pallidum antibody or human immunodeficiency virus antibody;
18. The clinical laboratory test results at the first screening (visit 1) and the baseline period (visit 3) meet any of the following criteria: 1） Hemoglobin (Hgb) < 100g/l; 2） Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal value (ULN);3） Total bilirubin (TBIL) > 1.5 times the upper limit of normal value (except for the known Gilbert syndrome that meets the following requirements, that is, part of bilirubin indicates conjugated bilirubin < 35% of total bilirubin); 4） Triglyceride (TG) ≥ 5.7mmol/l; 5） Estimated glomerular filtration rate < 60 ml/min (estimated by CKD-EPI formula);
19. Regular drinking (weekly alcohol intake greater than 21 units (male) and 14 units / week (female) (1 unit = 360ml beer; 150ml wine; or 45ml Baijiu) within 3 months before screening, or unable to quit drinking during the test;
20. Those who lost more than 400 ml of blood / donated blood (except physiological blood loss of women) within 3 months before screening, received blood transfusion or used blood products, or planned to donate blood during the test or within 1 month (30 days) after the end of the test;
21. Patients with a history of needle fainting, blood fainting or inability to tolerate venipuncture；
22. History of drug abuse, drug abuse and addiction;
23. Patients with obvious mental disorders, epilepsy and other persons without behavioral ability or cognitive ability;
24. History of malignant tumor or currently suffering from any malignant tumor;
25. Female subjects in pregnancy, lactation or pregnancy test (blood HCG test) positive; And the subjects have fertility or sperm / egg donation plans during the test period and within 60 days after the end of the test and cannot take effective physical contraceptive measures (effective contraceptive measures include abstinence, sterilization, intrauterine device, or diaphragm method stipulated by local laws);
26. An intervention clinical trial has been completed or withdrawn within 1 month before screening, or is currently undergoing an intervention clinical trial, or has participated in other medical research activities, which is not suitable to participate in this trial according to the judgment of the researcher;
27. The subjects may not be able to complete the test for other reasons or the researchers think they should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes of HbA1c compared with baseline at 12 weeks | 12 weeks
  Changes of HbA1c in each dose group compared with baseline at 12 weeks of treatment

SECONDARY OUTCOMES:
Changes of HbA1c compared with baseline at 8 weeks | 8 weeks
  Changes of HbA1c in each dose group compared with baseline at 8 weeks of treatment
Changes of maximum blood glucose increase (0-180min) after breakfast compared with baseline at 12 weeks | 12 weeks
  Changes of maximum blood glucose increase (0-180min) after breakfast in each dose group compared with baseline at 12 weeks of treatment
Proportion of subjects with HbA1c ≤ 7% | 8 weeks，12 weeks
Proportion of subjects with HbA1c ≤ 6.5% | 8 weeks，12 weeks
Changes of blood glucose at 2h after breakfast compared with baseline | 12 weeks
Changes of insulin at 2h after breakfast compared with baseline | 12 weeks
Changes of C-peptide at 2h after breakfast compared with baseline | 12 weeks
Change of GLP-1 from baseline 2h after breakfast | 12 weeks
Change of GIP from baseline 2h after breakfast | 12 weeks
Change of mean fasting blood glucose from baseline | 12 weeks
Change of fasting blood glucose from baseline | 4 weeks，8 weeks，12 weeks
change of mean blood glucose value at 7 time points from baseline | 4 weeks，8 weeks，12 weeks
  Based on SMPG test,the change of mean blood glucose value at 7 time points from baseline
Changes of blood glucose at 2h after meal compared with baseline | 4 weeks，8 weeks，12 weeks
  Based on SMPG test,the Changes of blood glucose at 2h after meal (breakfast, lunch and dinner) compared with baseline
Changes in insulin resistance (HOMA-IR) from baseline | 12 weeks
Islet of Langerhans β Cellular function (HOMA- β） Change from baseline | 12 weeks
Blood drug concentration level | 4 weeks，8 weeks，12 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The Second Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The first hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Changsha Central Hospital, Changsha, Hunan
  - Chengdu Fifth People's Hospital, Chengdu, Sichan
  - Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang